CLINICAL TRIAL: NCT04363203
Title: VA Remote and Equitable Access to COVID-19 Healthcare Delivery (VA-REACH TRIAL)
Acronym: VA-REACH
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: concerns related to study drug
Sponsor: Salomeh Keyhani MD (U.S. Federal Agency)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Salomeh Keyhani MD, Professor of Medicine, University of California San Francisco, San Francisco VA Health Care System
Organization: San Francisco VA Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-30517
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: A 3-arm RCT to determine the efficacy of hydroxychloroquine or azithromycin compared to placebo in treating mild to moderate COVID-19 among Veterans in the outpatient setting.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible, consented patients will be randomized to a 1:1:1 treatment allocation, stratifying by age (<65, 65 or more) and region, and using randomly permutated blocks (block size of 3) within study site. Pharmacy is unblinded to study drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine: 2x200mg mg PO in the AM and 2x200mg PO in the PM on Day 1, followed by 200mg capsule in the AM and 200 mg in the PM on Days 2-5
  Interventions: Drug: Hydroxychloroquine
- Azithromycin (Active Comparator): Azithromycin: 2x250mg by mouth (PO) in the AM followed by 250mg PO every day on days 2-5
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): The pills packs for the 3 arms are identical.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine: 2x200mg mg .PO in the AM and 2x200mg PO in the PM on Day 1, followed by 200mg PO in the AM and 200 mg PO in the PM on Days 2-5.
  Arms: Hydroxychloroquine
Drug: Azithromycin — Azithromycin: 2x250mg by mouth (PO) in the AM on Day 1, followed by 250mg PO every day on Days 2-5.
  Arms: Azithromycin
Drug: Placebo oral tablet — Placebo in pill packs identical to study drugs
  Arms: Placebo

SUMMARY:
We propose a 3-arm RCT to determine the efficacy of hydroxychloroquine or azithromycin in treating mild to moderate COVID-19 among Veterans in the outpatient setting.

DETAILED DESCRIPTION:
SARS-CoV-2 is a novel coronavirus disease (COVID-19) that presents with fever, cough, and shortness of breath, and has a mortality rate of 2-4%. Outcomes are worse among the elderly and those with cardiovascular, respiratory, cancer and other co-morbidities. Several treatments are also emerging as promising therapeutic candidates, hydroxychloroquine and azithromycin - both available as generic pills and widely used for other indications - are potential options for treatment. A small randomized controlled trial (RCT) of hospitalized patients suggests chloroquine may be superior to placebo in promoting viral elimination and shortening disease course. Hydroxychloroquine is preferred to chloroquine in the U.S. A small non-randomized trial found azithromycin had a clinical benefit. When azithromycin and hydroxychloroquine are given together, they can cause cardiac side-effects that limit use in the outpatient setting. These drugs, however, have independent potential benefits against COVID-19 that require more rigorous study before either is considered standard of care. We propose a 3-arm RCT to determine the efficacy of hydroxychloroquine or azithromycin in treating mild to moderate COVID-19 among Veterans in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* willingness to take the study drug and ability to take oral medications
* able to be contacted by phone
* willing and able to give informed consent for participation in the study and agrees with its conduct and willing to email the study team a picture of their consent form

Exclusion Criteria:

Exclusion Criteria Based on National VA Data:

We will exclude individuals based on the following national VA data and chart review criteria:

* eGFR <30mL/min or dialysis
* aspartate transaminase (AST) or alanine transaminase (ALT) >5 times the upper limit of normal or cirrhosis in past 2 years
* hypersensitivity to chloroquine, hydroxychloroquine or other 4-aminoquinolines (e.g., amodiaquine), azithromycin or macrolides
* already taking hydroxychloroquine or azithromycin
* congestive heart failure with an ejection fraction (EF) <35% in past 2 years or hospitalization within past 6 months
* concomitant treatment with any QT prolonging drug
* history of cardiac arrest, ventricular fibrillation or ventricular tachycardia in past 5 years
* QT prolongation on any ECG in past 5 years
* potassium <3.5 meq/l in labs in past 2 years
* magnesium< 1/5 meq/l in any lab in past 2 years
* any patient who has not had follow-up with their primary care doctors in past 2 years
* any Veteran who cannot follow-up such as those with dementia, home based primary care or those with active psychosis documented in past 2 years
* G6PD deficiency

Exclusions Based on Baseline Interview:

* any female who is breastfeeding or pregnant or planning to become pregnant.
* any Veteran who receives most of their care in non-VA settings
* Veteran enrolled in another COVID Trial
* Veteran received a prescription for azithromycin and hydroxychloroquine
* Veteran allergic to azithromycin and or hydroxychloroquine
* Veteran receiving QT prolonging drugs from non-VA pharmacy

Min Age: 216 Months | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Days to resolution of cough, fever and shortness of breath | 30-days

SECONDARY OUTCOMES:
Days to resolution of all COVID-19 symptoms | 30-days
All cause hospitalization | 30-days
All cause mortality | 30-days
COVID-19 specific mortality | 30-days
COVID-19 specific hospitalization | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Salomeh Keyhani, MD MPH, Principal Investigator — San Francisco VA/University of California, San Francisco
Locations (1):
- San Francisco VA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keyhani S, Kelly JD, Bent S, Boscardin WJ, Shlipak MG, Leonard S, Abraham A, Lum E, Lau N, Austin C, Oldenburg CE, Zillich A, Lopez L, Zhang Y, Lietman T, Bravata DM. A telehealth-based randomized controlled trial: A model for outpatient trials of off-label medications during the COVID-19 pandemic. Clin Trials. 2021 Aug;18(4):514-517. doi: 10.1177/17407745211011577. Epub 2021 May 20. PMID 34011199